CLINICAL TRIAL: NCT01033422
Title: A Phase 2, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Daily CF101 Administered Orally in Subjects With Elevated Intraocular Pressure
Brief Title: Safety and Efficacy of Daily CF101 Administered Orally in Subjects With Elevated Intraocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-231GL
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Ocular Hypertension; Glaucoma
Keywords: Glaucoma; Ocular hypertension; Intraocular hypertension
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CF101 1mg (Experimental): CF101 1mg orally q12 hours
  Interventions: Drug: CF101
- Placebo (Placebo Comparator): matching placebo orally q12 hours
  Interventions: Drug: Placebo for
- CF101 2mg (Experimental): CF101 2mg orally q12 hours
  Interventions: Drug: CF101

INTERVENTIONS:
Drug: CF101 — CF101 1 or 2 mg tablets orally every 12 hours for 16 weeks
  Other Names: IB-MECA
  Arms: CF101 1mg; CF101 2mg
Drug: Placebo for — Matching placebo tablets orally every 12 hours for 16 weeks
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This study will test the hypothesis that CF101, administered orally, will reduce intraocular pressure in patients with ocular hypertension and/or glaucoma. Eligible patients with elevated intraocular pressure will be evaluated and treated by ophthalmologist investigators, and will receive either CF101 pills or placebo (dummy) pills twice daily for 16 weeks. Ocular pressure, visual fields, and other aspects of safety and effectiveness will be monitored on a regular basis.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-masked, placebo-controlled, parallel-group study in adult males and females, aged 18 years and over, with a diagnosis of glaucoma or ocular hypertension.

This trial will be performed in 2 segments. In Segment 1, subjects will be randomized to receive either CF101 1.0 mg, or matching placebo, given orally every 12 hours for 16 weeks. Segment 1 will enroll approximately 44 subjects, randomized in a 3:1 ratio to CF101 1.0 mg or to placebo. At the conclusion of Segment 1, a Data Review Committee (DRC) will review safety and efficacy data and advise on progression of the trial to Segment 2. Segment 2 will enroll up to approximately 44 subjects randomized in a 3:1 ratio to CF101 2.0 mg 3:1 ratio to receive with CF101 2.0 mg, or matching placebo, given orally every 12 hours for 16 weeks.

At a Screening Visit (Visit 1, performed within 4 weeks prior to Baseline), subjects who provide written informed consent will have screening procedures performed, including complete medical, ophthalmologic, and medication histories; physical examination; vital signs and weight; electrocardiogram (ECG); ophthalmologic examination; tonometry; visual field (VF) assessment; corneal pachymetry; evaluation of inclusion and exclusion criteria; safety laboratory tests; serum pregnancy test for all females of child-bearing potential; and collection of concomitant medication information.

Subjects who successfully qualify will be randomized at Baseline (Visit 2) to their assigned medication (CF101 or matching placebo) to be taken orally every 12 hours for 16 weeks. Subjects will return for assessments and a new supply of study medication at Weeks 2, 4, 8, 12, and for final assessment and discharge at Week 16. A safety telephone call will be made at Week 18.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age and over;
2. Ocular hypertension or open-angle glaucoma in at least 1 eye, diagnosed as any of the following:

   1. Untreated ocular hypertension without glaucomatous anatomic or VF changes; or
   2. Glaucoma diagnosed within the past 2 months but untreated;
   3. Previously treated glaucoma, provided that previous medication treatment has been inefficacious and/or intolerable, and has therefore been discontinued at least 3 weeks prior to Baseline; or
   4. Currently treated glaucoma with inadequate IOP control, meaning that IOP remains above target pressure as judged by the Investigator despite ≥3 weeks of treatment with a standard topical regimen (for guidance, the European Glaucoma Society defines "target pressure" as follows: "In most cases a peak IOP = 8 mm - 15 mmHg on a diurnal curve, or 30% IOP reduction from baseline");
3. In subjects receiving a standard topical treatment regimen (per 2.d. above), the regimen and dose have not changed within 3 weeks of Screening, and are expected to remain stable throughout the treatment period;
4. At both Screening and Baseline, IOP in at least 1 eye ("candidate" eye) is >21 mmHg at 0800-1000 hours and >21 mmHg in at least 1 measurement at least 3 hours following the first;
5. Corneal thickness between 500 and 580 microns in both eyes;
6. Corrected visual acuity +0.18 logMAR or better by Early Treatment Diabetic Retinopathy Study (ETDRS) methodology in the candidate eye (equivalent to 20/30);
7. Females of child-bearing potential must have a negative urine pregnancy test at screening and throughout the study, to be eligible for, and continue participation in, the study;
8. Females of child-bearing potential must be willing to use 2 methods of contraception deemed adequate by the Investigator (eg, oral contraceptive pills plus a barrier method) to be eligible for, and continue participation in, the study;
9. Ability to complete the study in compliance with the protocol; and
10. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. IOP >32 mmHg in either eye;
2. History of angle-closure glaucoma;
3. Anatomically narrow angles in either eye (ie, ≥75% of the circumference of the angle must be ≥Grade 2 by Shaffer criteria );
4. In subjects with glaucoma, advanced VF defect in either eye, determined on reliable testing using the Humphrey Full-Threshold Algorithm for the Glaucoma Hemifield Test, defined as either:

   1. Mean deviation worse than -16 dB, or
   2. Threat to fixation (sensitivity 10 dB or worse affecting either or both test points closest to the point of fixation in the upper hemifield and at either or both the corresponding test points in the lower hemifield);
5. In subjects with ocular hypertension, a score of >12 points on The Ocular Hypertension Treatment Study Group and European Glaucoma Prevention Study Group Primary Open-Angle Glaucoma Risk Table;
6. Documented disc hemorrhage within the past 5 years in either eye;
7. Secondary cause of IOP elevation;
8. Glaucoma laser treatment in candidate eye within the past 3 months;
9. Clinically significant ocular trauma to candidate eye within the past 6 months;
10. Any major ocular surgery in the past, including keratorefractive surgery, in candidate eye, except for uncomplicated cataract surgery performed greater than 6 months prior to Screening;
11. Astigmatism >3 diopters in either eye;
12. Clinically significant acute or chronic ocular disease (eg, corneal edema, uveitis, severe keratoconjunctivitis sicca, active ocular infection, active herpes simplex keratitis, blepharitis, or acute conjunctivitis) that might interfere with the study;
13. Concomitant contact lens use;
14. Concomitant use of systemic medication that may affect IOP (eg, beta blockers, corticosteroids, calcium channel blockers, ACE inhibitors, or carbonic anhydrase inhibitors); however, systemic antihypertensive medications are allowed providing that the dose and regimen have been stable for at least 3 months prior to Screening and are expected to remain stable throughout the trial;
15. Any abnormality preventing reliable applanation tonometry;
16. Presence of uncontrolled asthma;
17. Presence of uncontrolled arterial hypertension or symptomatic hypotension;
18. Significant cardiac arrhythmia or conduction block, congestive heart failure (New York Heart Association Class 3-4), or any other evidence of clinically significant heart disease or clinically significant findings on screening ECG;
19. Hemoglobin level <9.0 gm/L, at screening;
20. Platelet count <125,000/mm3, at screening;
21. White blood cell count <3500/mm3, at screening;
22. Serum creatinine level greater than 1.5 times the laboratory's upper limit of normal (ULN), at screening;
23. Liver aminotransferase levels greater than 2 times the laboratory's ULN, at screening;
24. Known or suspected immunodeficiency or human immunodeficiency virus positivity;
25. Known infection with hepatitis B or C;
26. Pregnancy, planned pregnancy, lactation, or inadequate contraception as judged by the Investigator;
27. Previous receipt of CF101;
28. History of malignancy within the past 5 years (excluding basal cell carcinoma of the skin and ≤3 cutaneous squamous cell carcinomas, all of which have been completely excised);
29. Active drug or alcohol dependence;
30. Significant acute or chronic medical, ophthalmic, neurologic, or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study;
31. Participation in another investigational drug or vaccine trial concurrently or within 30 days; or
32. Other conditions which would confound the study evaluations or endanger the safety of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-10; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma
Locations (3):
- Bulgaria (2):
  - Specialized Hospital for Active Treatment for Eye Diseases "Zrenie", Sofia
  - University Multiprofile Hospital for Active Treatment "Tsaritsa Yoanna - ISUL", Sofia
- Bnei Zion Medical Center, Haifa, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- CF101 1mg: CF101 1 mg orally q12 hours
  CF101: CF101 1 mg tablets orally every 12 hours for 16 weeks
- CF101 2mg: CF101 2 mg orally q12 hours
  CF101: CF101 2 mg tablets orally every 12 hours for 16 weeks
Period: Overall Study
Arm/Group | CF101 1mg | CF101 2mg | Placebo
Started | 34 | 32 | 23
Completed | 33 | 28 | 22
Not Completed | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF101 1mg | CF101 2mg | Placebo | Total
Number analyzed (Participants) | 34 | 32 | 23 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.08 (9.513) | 55.51 (13.827) | 56.26 (11.303) | 56.83 (11.828)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 20 | 73
  Male | 9 | 4 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure in mmHg
Description: The mean of the IOP measurements obtained at week 16
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Intraocular Pressure in mmHg
Arm/Group | CF101 1mg | CF101 2mg | Placebo
Number analyzed (Participants) | 33 | 32 | 23
Intraocular Pressure in mmHg | 19.01 (3.001) | 19.84 (7.662) | 18.95 (4.237)

2. Secondary Outcome: Safety of CF 101
Description: To tabulate and enter the frequency (number) of adverse events during the treatment period of CF 101, by treatment arm.
Time Frame: 16 weeks
Measure: Number; unit: Number of events
Arm/Group | CF101 1mg | CF101 2mg | Placebo
Number analyzed (Participants) | 34 | 32 | 23
Number of events | 7 | 11 | 10

ADVERSE EVENTS:
Arm/Group | CF101 1mg | CF101 2mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/32 | 0/23
Other Adverse Events (participants affected / at risk) | 4/34 | 4/32 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 1mg (N=34) | CF101 2mg (N=32) | Placebo (N=23)
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 1mg (N=34) | CF101 2mg (N=32) | Placebo (N=23)
Any (Eye disorders) | 0 | 1 | 2
Any (Gastrointestinal disorders) | 0 | 1 | 2
Any (Infections and infestations) | 4 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No